CLINICAL TRIAL: NCT04350645
Title: Role of Prophylactic Tranexamic Acid in Reducing Blood Loss During Elective Caesarean Section for Placenta Praevia Major: A Randomized Controlled Study
Brief Title: Role of Prophylactic Tranexamic Acid in Reducing Blood Loss During Elective Caesarean Section for Placenta Praevia Major
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Chew Kah Teik, Clinical lecturer and gynaecologist, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UKM PPI/1118/JEP-2019-846
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Hemorrhage From Placenta Previa, With Delivery
MeSH Terms: interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid group (Active Comparator): Tranexamic acid group will receive 1g slow bolus of tranexamic acid over 2 minutes at least 5 minutes before skin incision (at the end of spinal/general anaesthesia)
  Interventions: Drug: Tranexamic acid injection
- Control group (Placebo Comparator): The placebo group will receive normal saline 0.9% (same amount as the tranexamic acid)
  Interventions: Drug: Normal Saline 0.9%

INTERVENTIONS:
Drug: Tranexamic acid injection — 1g slow bolus of tranexamic acid over 2 minutes
  Arms: Tranexamic acid group
Drug: Normal Saline 0.9% — 10mls normal saline 0.9% over 2 minutes
  Arms: Control group

SUMMARY:
Prophylactic tranexamic acid will reduce blood loss during Caesarean section for placenta praevia

DETAILED DESCRIPTION:
Tranexamic acid is a promising agent, easy to administer, cheap, and can be added to the other routine management in hospitals deliveries. This study aims to document the efficacy of intravenous tranexamic acid in reducing blood loss during and after caesarean section in placenta praevia major patients and to assess the Hb and platelet change after its administration.

General objective:

To investigate the effect of prophylactic IV tranexamic acid in reducing blood loss during Caesarean section for placenta praevia major

Specific objectives:

1. To evaluate the effect of prophylactic IV tranexamic acid in reducing blood loss during Caesarean section up to 2 hours after Caesarean section.
2. To evaluate the drop in Haemoglobin level postoperatively with the use of prophylactic IV tranexamic acid for Caesarean section for PP major
3. To examine the effect of tranexamic acid on platelet level for caesarean section for PP major
4. To observe the side effects of tranexamic acid

This study will be conducted at University Kebangsaan Malaysia Medical Centre (UKMMC). Patients who meet the inclusion criteria will be invited to participate in the study. Patient will be given the information sheet regarding the study and consent will be taken if agreeable to participate. Patients' demographic data will be recorded.

Patients will be classified randomly into two groups using a computer-generated randomization system (Microsoft Office Excel). The list of randomization will be concealed and numbered on sealed opaque envelopes. Each number will be given a readily prepared 10ml syringe of colourless solution, which could either contain the tranexamic acid or placebo.

Each patient will be assigned a serial identification number. The data will be analysed using the Statistical Package for Social Sciences (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* all placenta previa major pregnant women

Exclusion Criteria:

1. Any cardiac disorder or liver disease
2. Patient on anticoagulant therapy
3. History of allergy to tranexamic acid
4. Any contraindication for tranexamic acid

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2021-12-23 (Estimated); Study Completion 2021-12-23 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of prophylactic IV tranexamic acid in amount of blood loss during Caesarean section in placenta previa major | 24 hours
  Amount of blood loss in mls
To evaluate the effect of prophylactic IV tranexamic acid in the changes of haemoglobin during Caesarean section in placenta previa major | 24 hours
  changes of haemoglobin level

SECONDARY OUTCOMES:
To evaluate the side effects of tranexamic acid | one week
  platelet count

CONTACTS AND LOCATIONS:
Overall Officials: Kah Teik Chew, Principal Investigator — UKM Medical Centre
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur, Malaysia